CLINICAL TRIAL: NCT03568097
Title: Phased Avelumab Combined With Chemotherapy as First-line Treatment for Patients With Advanced Small-cell Lung Cancer (SCLC)
Brief Title: Immunotherapy in Combination With Chemotherapy in Small-cell Lung Cancer
Acronym: PAVE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hellenic Cooperative Oncology Group (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE1/17; 2017-004784-12 (EudraCT Number)
Record Dates: First submitted 2018-05-30; First posted 2018-06-26 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab + Standard 1st line Chemotherapy (Experimental): Administration of cisplatin or carboplatin + etoposide every 3 weeks with phased avelumab administered every 2 weeks until disease progression.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — 10 mg/kg will be given as intravenous infusion (IV) every two weeks (q 2 weeks) until disease progression.
  Other Names: Bavencio

SUMMARY:
PAVE(Phased Avelumab combined with chemotherapy as first-line treatment for patients with advanced small-cell lung cancer) is a Greek, investigator- initiated, single arm open- label phase II study of Avelumab in combination with cisplatin or carboplatin/ etoposide.

The study will include an initial safety run-in, open-label, singlearm part (Part 1), and the actual phase II study (Part 2). The total number of patients will not change (the safety run-in patients will be included in the final total number of participants). The safety run-in period will not alter the total study timelines, as phase II accrual will follow immediately after the safety run-in.

DETAILED DESCRIPTION:
Advanced small cell lung cancer (SCLC) remains a disease with dismal prognosis and new therapeutics are urgently needed. SCLC is notably chemosensitive and first-line chemotherapy with platinum analogs and etoposide is associated with high rates of initial objective responses that unfortunately do not last long.

The primary endpoint for study design is 1-year PFS rate, where according to RECIST v1.1 PFS is determined as the time from the date of study entry to the date of progression, death from any cause or date of last contact.Secondary End Point is the evaluation of efficacy of the study treatment in terms of Overall Survival (OS), Best Overall Response (BOR), Objective Response Rate (ORR) and Duration of Response (DOR).

Evaluation of the safety of the study treatment by assessing Treatment-Emergent Adverse Events (TEAEs).

Evaluation of the Quality of Life of patients receiving the study the study treatment. Evaluation of potential biomarkers on fresh or archival sample,of formalin-fixed paraffin embedded tumor tissue block or a minimum of 10 unstained tumor tissue sections. Moreover 10 ml of EDTA-stored blood sample will be collected as well.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female patients aged more than or equal to (≥) 18 years
* With Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1 at trial entry
* At least 1 measurable tumor lesion by RECIST 1.1
* With histologically confirmed metastatic (Stage IV) small cell lung cancer (SCLC)
* Patients must not have received any previous systemic treatment for small cell lung cancer
* Patients must have an estimated life expectancy of more than 12 weeks
* Patients must have an available recently-obtained, formalin-fixed, paraffin-embedded (FFPE) tissue sample containing tumor (biopsy preferably within 6 months) or a minimum number of 10 unstained slides, suitable for PD-L1 expression assessment.

Exclusion Criteria:

* Patients with brain metastases are excluded, except those with brain metastases that have been treated with surgery or radiation and are clinically stable for at least 2 weeks prior to registration.
* Prior therapy with any antibody or drug targeting T cell co-regulatory proteins, concurrent anticancer treatment, or immunosuppressive agents
* Patients on current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)."
* Known severe hypersensitivity reactions to monoclonal antibodies, history of anaphylaxis, or uncontrolled asthma, and persisting toxicity related to prior therapy of Grade > 1 NCI-CTCAE v 4.03.
* Patients with active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent.
* Patients with prior organ transplantation including allogenic stem-cell transplantation are excluded.
* Patients with an active infection requiring systemic therapy are excluded.
* Patients with known history of testing positive for HIV or known acquired immunodeficiency syndrome are excluded.
* Also excluded are patients with Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
* Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines.
* Persisting toxicity related to prior therapy
* Other severe acute or chronic medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2018-09-16 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
1- year Progression Free Survival (PFS) Rate | Time from inclusion in the trial up to 12 months
  Efficacy of treatment for 1- year PFS according to RECIST v1.1

SECONDARY OUTCOMES:
Overall Survival Time (OS) | Time from inclusion in the trial until the date of death due to any cause, up to 30 months.
Best Overall Response (BOR). | Time from inclusion in the trial up to 30 months.
  Best Overall Response (BOR) according to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1). Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Stable disease (SD)=Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR.
Objective Response Rate (ORR). | Time from inclusion in the trial up to 30 months.
  Proportion of patients with CR or PR as the best overall response according to RECIST 1.1.
Duration of Response (DOR) according to RECIST Version 1.1 | Time from inclusion in the trial up to 30 months.
  DOR will be determined according to RECIST 1.1, defined for each subject with a confirmed response as the time from the date of the first assessment demonstrating a CR or PR to date of the first assessment demonstrating PD or death from any cause within 12 weeks after the last tumor assessment, whichever occurs first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Stable disease (SD)=Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. PD is defined as at least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03 | From the first dose of study drug treatment up to 90 days after the last dose of study drug administration
  TEAEs will be defined as the adverse events (AEs) that occur between first dose of study drug administration and 90 days after the last dose of study drug administration that were absent before treatment or that worsened relative to pretreatment state.
Change from baseline in European Quality Of Life 5-dimensions (EQ-5D-5L) Health Outcome Questionnaire | On Day 1 every 21 days for 18 weeks then monthly up to 30 months.
  The EQ-5D-5L Health Outcome Questionnaire is a measure of health status that provides a simple descriptive profile and a single index value. The EQ-5D-5L defines health in terms of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The 5 items are combined to generate health profiles. These profiles were converted to a continuous single index score using a one to one matching. The lowest possible score is -0.59 (unable to walk, unable to self-care, unable to do usual activities, extreme pain or discomfort, extreme anxiety or depression) and the highest is 1.00 (no problems in all 5 dimensions).
Change from baseline in European Organization for the Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) Global Health Status | On Day 1 every 21 days for 18 weeks then monthly up to 30 months.
  EORTC QLQ-C30 is a 30-question tool used to assess the overall quality of life (QoL) in cancer subjects. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, role, cognitive, emotional, social), and 9 symptom scales/items (Fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, financial impact. The EORTC QLQ-C30 GHS/QoL score ranges from 0 to 100; High score indicates better GHS/QoL. Score 0 represents: very poor physical condition and QoL. Score 100 represents: excellent overall physical condition and QoL.
Change from baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13) | On Day 1 every 21 days for 18 weeks then monthly up to 30 months.
  EORTC QLQ-LC13 consists of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy. The 13 questions comprises 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, neuropathy, alopecia, and medicine for pain). Score range: 0 (no burden of symptom domain or single symptom item) to 100 (highest burden of symptoms for symptom domains and single items).
Translational research | At baseline
  PD-L1 expression by immunohistochemistry on available tumour tissue collected from this study.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Linardou, MD, Principal Investigator — 1st Department on Medical Oncology, Metropolitan Hospital
Locations (6):
- Greece (6):
  - Attikon University Hospital, Chaïdári, Athens
  - Agii Anargiri Cancer Hospital, Nea Kifissia, Athens
  - Metropolitan Hospital, Neo Faliro, Athens
  - Patra University Hospital, Rio, Patra
  - Henry Dunant Hospital Center, Athens
  - Alexandra Hospital, Athens